CLINICAL TRIAL: NCT02876523
Title: Biliary Hilar Drainage Managed by Endoscopy
Acronym: HILARIUM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Other Study IDs: HILARIUM-IPC 2015-003
Record Dates: First submitted 2016-08-02; First posted 2016-08-23 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Hilar Biliary Strictures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with a hilar biliary stricture requiring a drainage: Drainage performed by endoscopy, echo-endoscopy or percutaneously

SUMMARY:
The management of hilar biliary strictures remains difficult. These strictures are classified in 4 types (I,II,III and IV). In palliative cases, an endoscopic drainage should be performed in types I and II while a percutaneous drainage is performed in type IV. There is controversy as to whether partial or complete liver drainage should be done. Furthermore there are no standards for drainage types (metallic stents, plastic stents). Morbidity remains high and a multistage procedure can be required.

This study aims at evaluating the clinical practices in the investigators' center in order to determine the key factors that contribute to the drainage success or failure.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Biliary strictures requiring a drainage

Exclusion Criteria:

* Contraindication to hilar biliary drainage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with a hilar biliary strictures requiring a drainage
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Efficacy evaluated by the need for re-interventions | up to 2 years
  Number of re-interventions
Efficacy evaluated by the need for re-hospitalization | up to 2 years
  Number of re-hospitalization
Efficacy evaluated by complete or partial liver drainage | up to 2 years
  realization of complete or partial liver drainage

SECONDARY OUTCOMES:
Toxicity: Occurrence of drainage complications (sepsis, hemorrhage) | up to 2 years
  Occurrence of drainage complications (sepsis, hemorrhage)

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli Calmettes, Marseille, Bouches du Rhone, France

IPD SHARING:
Plan to Share IPD: No